CLINICAL TRIAL: NCT06720402
Title: Increasing the Knowledge and Awareness Levels of Pediatricians and Family Physicians on Sun Protection Methods
Brief Title: Pediatricians and Family Physicians Knowledge and Awareness on Sun Protection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09.2024.255
Record Dates: First submitted 2024-05-17; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-05

CONDITIONS: Sun Protection; Skin Burn; Sunburn
Keywords: sun protection; children; pediatrician; family physician; preventative counseling
MeSH Terms: conditions — Paresthesia; Sunburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatricians (Active Comparator): The group which consist of pediatricians.
  Interventions: Behavioral: Sun protection knowledge
- Family physicians (Active Comparator): The group which consist of family physicians.
  Interventions: Behavioral: Sun protection knowledge

INTERVENTIONS:
Behavioral: Sun protection knowledge — To increase knowledge and awareness about sun protection methods, a presentation will be implented to pediatricians and family physicians.

SUMMARY:
Sunlight has very important effects on the body. In addition to its positive effects such as regulation of circadian rhythm, synthesis of vitamin D and regulation of mood, it also has negative effects on the skin such as sunburn, hyperpigmentation, photoaging and skin cancer formation. These negative effects are known to be caused by ultraviolet (UV) (10 to 400 nm) rays of sunlight.

It is known that skin cancers such as melanoma, basal cell carcinoma and squamous cell carcinoma may develop in adults as a result of excessive exposure to UV rays. It has been shown that the development of skin cancer is rare in childhood.

Although skin cancers are not common in the pediatric age group, exposure to UV rays is higher than in adults. It is known that this cumulative exposure that develops over time may lead to the development of skin cancer in later ages. Therefore, it is argued that effective protection from UV rays is important in the pediatric age group. Guidelines emphasize the importance of preventive counseling in early childhood for reasons such as high sun exposure in the pediatric age group, increase in cumulative exposure with advancing age, prevention of the known adverse effects of sun rays with simple precautions, application of sun protection trainings given to the child for the rest of his/her life and thus decreasing the incidence of skin cancers. The World Health Organization and the American Academy of Pediatrics emphasize the following 5 basic points about reducing UV exposure in early childhood:

* Avoid going outside between 10.00-15.00 when the sun is at its peak,
* Usage of broad spectrum sunscreen children over 6 months,
* Using a hat, clothing that fully protects the body, sunglasses, umbrellas when going outside,
* When spending time outdoors, spend more time in shaded areas,
* Avoidance of indoor tanning.

In this sense, it is of critical importance that all physicians have the necessary knowledge and equipment to provide preventive counseling on the negative effects of sunlight on the skin and cancer development.

In this study, it is aimed to investigate the knowledge levels of Pediatricians and Family Physicians about sun protection and to increase their knowledge and awareness levels about sun protection in order to provide preventive counseling for the pediatric age group and their families.

DETAILED DESCRIPTION:
Sunlight has very important effects on the body. In addition to its positive effects such as regulation of circadian rhythm, synthesis of vitamin D and regulation of mood, it also has negative effects on the skin such as sunburn, hyperpigmentation, photoaging and skin cancer formation. These negative effects are known to be caused by ultraviolet (UV) (10 to 400 nm) rays of sunlight.

UV waves reaching the Earth are divided into three as Ultraviolet A (UV-A), Ultraviolet B (UV-B) and Ultraviolet C (UV-C). Approximately 95% of the UV rays reaching the Earth's surface are UV-A (320 to 400 nm). UV-A is known to contribute to photoaging, play an important role in hyperpigmentation and cause the development of skin cancer. UV-B (290 to 320 nm) constitutes 5% of UV radiation and contains the most biologically active wavelengths. UV-B is known to cause sunburn, inflammation, hyperpigmentation and skin cancer development. It is known that UV-C (200 to 290 nm) cannot reach the earth due to the ozone layer.

It is known that skin cancers such as melanoma, basal cell carcinoma and squamous cell carcinoma may develop in adults as a result of excessive exposure to UV rays. It has been shown that the development of skin cancer is rarer in childhood. It has been found that approximately 324 thousand patients worldwide are diagnosed with melanoma and 1.2 million patients are diagnosed with non-melanoma skin cancer each year. In Turkey, according to the latest data, 1477 patients were diagnosed with melanoma and 20,220 patients were diagnosed with non-melanoma skin cancer. According to Fitzpatrick skin classification, studies have found that the risk of cancer development is higher in light-skinned skin, while the risk of cancer development is lower in dark-skinned skin.

Although skin cancers are not common in the pediatric age group, exposure to UV rays is higher than in adults. It is known that this cumulative exposure that develops over time may lead to the development of skin cancer in later ages. Therefore, it is argued that effective protection from UV rays is important in the pediatric age group. Guidelines emphasize the importance of preventive counseling in early childhood for reasons such as high sun exposure in the pediatric age group, increase in cumulative exposure with advancing age, prevention of the known adverse effects of sun rays with simple precautions, application of sun protection trainings given to the child for the rest of his/her life and thus decreasing the incidence of skin cancers. The World Health Organization and the American Academy of Pediatrics emphasize the following 5 basic points about reducing UV exposure in early childhood:

* Avoid going outside between 10.00-15.00 when the sun is at its peak,
* Usage of broad spectrum sunscreen children over 6 months,
* Using a hat, clothing that fully protects the body, sunglasses, umbrellas when going outside,
* When spending time outdoors, spend more time in shaded areas,
* Avoidance of indoor tanning.

In this sense, it is of critical importance that all physicians have the necessary knowledge and equipment to provide preventive counseling on the negative effects of sunlight on the skin and cancer development. In our country, it is known that Family Physicians working in the first step and Pediatricians working in fields take part in the provision of early childhood preventive health services. However, it is seen in the literature that both Pediatricians and Family Physicians do not have sufficient knowledge about sun protection methods and preventive counseling on this subject needs to be emphasized more in medical education.

In this study, it is aimed to investigate the knowledge levels of Pediatricians and Family Physicians about sun protection and to increase their knowledge and awareness levels about sun protection in order to provide preventive counseling for the pediatric age group and their families.

All participants will participate in a presentation about sun protection. Also motivational interviewing methods organized by a team of professionals in the field will be used in the planning and implementation of the presentation.

The training will be prepared as a presentation. The presentation will last at least 30 minutes. It will be conducted using Microsoft Powerpoint presentation, face to face as a group and motivational interviewing techniques will be implemented during session. Presentation will include the current recommendations of the American Academy of Pediatrics and the World Health Organization and will be prepared using appropriate data and visuals. The training content consists of 4 main topics:

1. Purpose of the training program,
2. Skin properties and functions,
3. Sun rays, positive and negative effects of sun rays and skin diseases caused by sun rays,
4. The importance of providing preventive counseling on sun protection and information on sun protection methods outlined by the American Academy of Pediatrics and the World Health Organization.

The knowledge level will be assessed by Skin Cancer and Sun Knowledge scale immediately before and after the program and at the 3th month.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics residents and specialists
* Family medicine residents and specialists
* Family physicians working at family medicine centers

Exclusion Criteria:

* Medical students
* Physicians working at other fields
* Attendants who have skin cancer history at him/herself and in family

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Sun protection methods | Baseline and up to 3rd months.
  A presentation consisting of WHO and AAP recommendations will be given and to measure the increase in knowledge and awareness of healthcare professionals, the Skin Cancer and Sun Knowledge scale will be measured at baseline, at the end of the presentation and after 3 months. An increase in the total score indicates an increase in knowledge and awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Day AK, Wilson C, Roberts RM, Hutchinson AD. The Skin Cancer and Sun Knowledge (SCSK) Scale: Validity, Reliability, and Relationship to Sun-Related Behaviors Among Young Western Adults. Health Educ Behav. 2014 Aug;41(4):440-8. doi: 10.1177/1090198114529129. Epub 2014 Apr 10. PMID 24722215
- [Result] Green AC, Wallingford SC, McBride P. Childhood exposure to ultraviolet radiation and harmful skin effects: epidemiological evidence. Prog Biophys Mol Biol. 2011 Dec;107(3):349-55. doi: 10.1016/j.pbiomolbio.2011.08.010. Epub 2011 Sep 3. PMID 21907230
- [Result] Araujo FM, Carmo JAD, Cunha LD, Martins IML, Gon ADS, Caldeira AP. Development and validation of an instrument to assess the knowledge of general practitioners and pediatricians about photoprotection and solar radiation. An Bras Dermatol. 2019 Sep-Oct;94(5):532-541. doi: 10.1016/j.abd.2019.09.011. Epub 2019 Sep 30. PMID 31777353
- [Result] Balk SJ. Sun Protection. Pediatr Rev. 2023 Apr 1;44(4):236-239. doi: 10.1542/pir.2022-005545. No abstract available. PMID 37002351
- See also: EPA Recommendations — https://www.epa.gov/radtown/ultraviolet-uv-radiation-and-sun-exposure
- See also: American Academy of Dermatology Recommendations — https://www.aad.org/media/stats-sunscreen
- See also: FDA Sunscreen Recommendations — https://www.fda.gov/drugs/understanding-over-counter-medicines/sunscreen-how-help-protect-your-skin-sun
- See also: Related Info — https://www.healthychildren.org/English/safety-prevention/at-play/Pages/Sun-Safety.aspx